CLINICAL TRIAL: NCT00859157
Title: Tumescent Mastectomy: A Prospective Comparison to Standard Mastectomy Technique
Brief Title: Pain After Tumescent Mastectomy or Standard Mastectomy in Women With Stage I, Stage II, or Stage III Breast Cancer
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 246600; UCD-CCSO001; 200816282; CDR0000633754 (Other: UC Davis)
Record Dates: First submitted 2009-03-07; First posted 2009-03-10 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Breast Cancer; Pain; Perioperative/Postoperative Complications
Keywords: perioperative/postoperative complications; pain; ductal breast carcinoma in situ; invasive ductal breast carcinoma; invasive lobular breast carcinoma; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms; Pain; Postoperative Complications; Carcinoma, Intraductal, Noninfiltrating; Carcinoma, Ductal, Breast; Carcinoma, Lobular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: Patients undergo standard mastectomy.
  Interventions: Procedure: therapeutic conventional surgery
- Group 2: Patients undergo tumescent mastectomy.
  Interventions: Procedure: therapeutic conventional surgery

INTERVENTIONS:
Procedure: therapeutic conventional surgery — Patients undergo tumescent or standard mastectomy

SUMMARY:
RATIONALE: New surgery techniques may lessen pain after breast surgery. It is not yet known whether tumescent mastectomy or standard mastectomy results in less pain in women with breast cancer.

PURPOSE: This clinical trial is studying pain after tumescent mastectomy compared with pain after standard mastectomy in women with stage I, stage II, or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare post-operative pain after tumescent vs standard mastectomy in women with stage I-III breast cancer.

Secondary

* To compare the total time of operation from incision to completion of wound closure.
* To compare the time of operation from first incision to completion of skin flaps.
* To compare the total estimated blood loss.
* To compare the number of days the Jackson-Pratt drain is left in place under skin flaps with wound drainage > 30 mL/24 hours.
* To compare the incidence of wound complications such as skin necrosis, hematoma, cellulitis, abscess, and seroma between groups.

OUTLINE: Patients are grouped according to which surgeon provided their evaluation and treatment recommendations.

* Group 1: Patients undergo standard mastectomy.
* Group 2: Patients undergo tumescent mastectomy. All patients receive standardized post-operative pain management comprising morphine sulfate for analgesia or an equivalent dose of hydromorphone hydrochloride for 24 hours following surgery. Patients then receive 1-2 oral acetaminophen/oxycodone hydrochloride combination tablets (or a comparable amount of another narcotic/acetaminophen combination) every 6 hours as needed. Pain is assessed using the Short-form McGill Pain Questionnaire (SF-MPQ).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of 1 of the following:

  * Invasive (ductal or lobular) breast cancer
  * In situ (ductal) breast cancer
* Stage 0-III disease
* Localized disease
* Candidate for curative mastectomy and selected mastectomy or modified radical mastectomy for surgical option of treatment at the University of California Davis Medical Center
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* WBC ≥ 1,500/mm^3
* Platelet count ≥ 90,000/mm^3
* PT/PTT ≤ upper limit of normal (ULN)
* Creatinine ≤ 1.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* No NYHA cardiac disease class III-IV
* Cancer survivors must have undergone potentially curative therapy for all prior malignancies with no evidence of prior malignancy within the last 5 years, except for effectively treated basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix treated by surgery alone, or lobular carcinoma in situ of the breast treated by surgery alone
* Body Mass Index ≤ 40

PRIOR CONCURRENT THERAPY:

* No prior major breast surgery, including breast augmentation or reduction surgery
* No preoperative chemotherapy or radiotherapy
* No concurrent immediate breast reconstruction
* No concurrent bilateral mastectomy
* No concurrent narcotic pain medication

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (age 18 or more) women with histologic diagnosis of stage 0, I, II, III breast cancer undergoing mastectomy.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2008-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Post-operative pain at 1 and at 7-10 days after mastectomy | 7-10 days

SECONDARY OUTCOMES:
Number of acetaminophen/oxycodone tablets taken | 7-10 days after surgery
Total time of operation from breast incision to completion of wound closure | Day of surgery
Time of operation from first incision to completion of both superior and inferior skin flaps | Day of surgery
Estimated blood loss | Day of surgery
Number of days the Jackson-Pratt drain is left in place with wound drainage > 30 mL/24 hours | 7-10 days after surgery
Wound complications (skin necrosis, hematoma, cellulitis, abscess, and seroma) occurring up to and 10 days post-operatively | Up to 10 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Steve R. Martinez, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Cancer Center, Sacramento, California, United States